CLINICAL TRIAL: NCT02032121
Title: Vascular Endothelial Inflammation and Dysfunction in Pediatric Long-term Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Tracie L. Miller, MD, Professor of Pediatrics, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20070584
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Cancer Survivor; Pediatric Cancer
Keywords: Cancer survivors; Long-term cancer survivor
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection; Carotid Intima-Media Thickness; Bone Density

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention procedures (Experimental): All the procedures will be completed for every subject
  Interventions: Procedure: Blood specimen; Procedure: Echocardiography

INTERVENTIONS:
Procedure: Blood specimen
Procedure: Echocardiography
  Other Names: Flow mediated vasodilation; Carotid intimal media thickness; Bone Mineral Density

SUMMARY:
Survivors of childhood cancer have an increased risk of death from cardiovascular disease due to both the therapies they received while undergoing treatment and diet and lifestyle factors. The nature of cardiovascular risk and the interaction between treatment affects and cardiovascular risk factors is unknown. We propose to study vascular inflammatory markers as well as measure of blood vessel stiffness (both of which are predictive of early heart disease) in 100 pediatric cancer survivors and 100 control children. Characterization of vascular inflammation and stiffness in long-term survivors will allow for the development of future interventions to decrease inflammation through both pharmacologic and lifestyle modifications.

ELIGIBILITY:
Inclusion Criteria:

* 6-30 years of age
* 2 years from the completion of therapy for cancer
* free of active disease

Exclusion Criteria:

* <6 or > 30 years of age
* current cancer treatment or inside of 2 years post treatment
* Active disease/infection

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2007-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Vascular Inflammation | single time point at initial visit
  All study procedures to assess vascular inflammation will be assessed through specimen sample collection and through procedures such as (echocardiograph)

CONTACTS AND LOCATIONS:
Overall Officials: Tracie L Miller, MD, SM, Principal Investigator — University of Miami
Locations (1):
- University of Miami, MIller School of Medicine, Miami, Florida, United States